CLINICAL TRIAL: NCT01336296
Title: A 12-month, Prospective, Randomized, Dual Center, Open Label Pilot Study to Evaluate the Safety and Efficacy of Myfortic® (Mycophenolic Acid) Loading Regimens in Combination With Thymoglobulin® [Anti-thymocyte Globulin (Rabbit)] or Simulect® (Basiliximab) Induction and Prograf® (Tacrolimus) in Early Corticosteroid Withdrawal
Brief Title: Evaluate Effects and Safety of Pre-load Myfortic® in Transplant Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Cincinnati (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Adele Rike-Shields, PharmD, University of Cincinnati
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Myfortic Preload
Record Dates: First submitted 2010-10-28; First posted 2011-04-15 (Estimated); Results first posted 2016-04-11 (Estimated); Last update posted 2016-08-02 (Estimated); Status verified 2016-07

CONDITIONS: Kidney Transplant Recipients
MeSH Terms: interventions — Mycophenolic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Myfortic preload (Active Comparator): Initiation of mycophenolic acid (Myfortic) 2 weeks prior to transplantation (with Simulect induction at time of transplant)
  Interventions: Drug: mycophenolic acid
- Myfortic standard (Active Comparator): mycophenolic acid (Myfortic) at time of transplant with Thymoglobulin induction
  Interventions: Drug: mycophenolic acid

INTERVENTIONS:
Drug: mycophenolic acid — Comparing mycophenolic acid 720mg orally twice daily starting 2 weeks prior to transplant to mycophenolic acid 720mg orally twice daily starting day of transplant.
  Other Names: Myfortic

SUMMARY:
This study is specifically designed to determine whether the initiation of Myfortic 2 weeks prior to transplantation will enhance the therapeutic efficacy of Simulect induction therapy in low to moderate risk patients. Specifically, the addition of Myfortic pretransplant to Simulect induction will be compared to standard Myfortic therapy with Thymoglobulin induction starting at the time of transplant in kidney transplant recipients.

ELIGIBILITY:
Inclusion Criteria:

* Patients capable of understanding the purposes and risks of the study.
* Patients who can give written informed consent, and who are willing and able to participate in the full course of the study.
* Women of childbearing potential must have a negative serum pregnancy test within the last 48 hours prior to receiving study medication.
* Women of childbearing potential must use two reliable forms of contraception simultaneously, unless they are status post bilateral tubal ligation, bilateral oophorectomy, or hysterectomy. Effective contraception must be used before beginning study drug therapy, for the duration of the study and for 6 weeks following completion of the study.

Exclusion Criteria:

* Patients who are recipients of a multiple organ transplant or if the patient previously received and organ transplant.
* Patients who are recipients of A-B-O incompatible transplants, all complement-dependent cytotoxicity (CDC) crossmatch positive transplants.
* Sensitized patients [most recent anti-Human Leukocyte Antigens (HLA) Class I panel reactive antibody (PRA) ≥ 25% by a CDC-based assay].
* Recipient or donor is known to be seropositive for hepatitis C virus (HCV) or B virus (HBV) except for hepatitis B surface antibody positive.
* Recipient or donor is known to be seropositive for human immunodeficiency virus (HIV).
* Patient has uncontrolled concomitant infection or any other unstable medical condition that could interfere with the study objectives.
* Patients with thrombocytopenia (<75,000/mm3 ), with an absolute neutrophil count of < 1,500/mm3); and/or leucopoenia (< 2,500/mm3), or anemia (hemoglobin < 6 g/dL) prior to study inclusion.
* Patient is taking or has been taking an investigational drug in the 30 days prior to transplant.
* Patient has a known hypersensitivity to tacrolimus, mycophenolate mofetil, enteric-coated mycophenolic acid, rabbit anti-thymocyte globulin, or corticosteroids.
* Patients with severe diarrhea or other gastrointestinal disorders that might interfere with their ability to absorb oral medication; diabetic patients with previously diagnosed diabetic gastroenteropathy, or patients with active peptic ulcer disease.
* Patient is receiving chronic steroid therapy at the time of transplant.
* Patients with a history of malignancy within the last five years, except for successfully excised squamous or basal cell carcinoma of the skin.
* Patient is pregnant or lactating, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by positive human Chorionic Gonadotropin (hCG) laboratory test.
* Patient has any form of substance abuse, psychiatric disorder or a condition that, in the opinion of the investigator, may invalidate communication with the investigator.
* Inability to cooperate or communicate with the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2010-09; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adele Shields, Pharm.D., Principal Investigator — University of Cincinnati
Locations (1):
- University of Cincinnati Medical Center, Cincinnati, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Myfortic Preload: Initiation of Myfortic 2 weeks prior to transplantation (with Simulect induction at time of transplant)
  mycophenolic acid: Comparing mycophenolic acid 720mg orally twice daily starting 2 weeks prior to transplant to mycophenolic acid 720mg orally twice daily starting day of transplant
- Myfortic Standard: Myfortic at time of transplant with Thymoglobulin induction
  mycophenolic acid: Comparing mycophenolic acid 720mg orally twice daily starting 2 weeks prior to transplant to mycophenolic acid 720mg orally twice daily starting day of transplant
Period: Overall Study
Arm/Group | Myfortic Preload | Myfortic Standard
Started | 40 | 21
Completed | 35 | 17
Not Completed | 5 | 4

BASELINE CHARACTERISTICS:
Population: Intent to treat
Groups:
- Total: Total of all reporting groups
Arm/Group | Myfortic Preload | Myfortic Standard | Total
Number analyzed (Participants) | 40 | 21 | 61
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.1 (15) | 55.8 (13.1) | 55.4 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 6 | 18
  Male | 28 | 15 | 43
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 2 | 7
  White | 35 | 19 | 54
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 40 | 21 | 61

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Biopsy-confirmed Acute Rejection by Banff '97 Criteria (Updated 2007) 3, 6 and 12 Months Post Transplant
Description: Incidence of biopsy-confirmed acute rejection by Banff '97 Criteria (updated 2007) post transplant. The acute form of T-cell mediated rejection is furthermore subclassified as follows. Since this is the most common form of rejection, it is useful to know:
  As with humoral rejection, there are both acute & chronic forms:
  The acute form of T-cell mediated rejection is furthermore subclassified as follows. Since this is the most common form of rejection, it is useful to know:
  Class IA: there is at least 25% of parenchymal showing interstitial infiltration and foci of moderate tubulitis (defined as a certain number of immune cells present in tubular cross-sections).
  Class IB: just like Class IA except there is more severe tubulitis.
  Class IIA: there is mild-to-moderate intimal arteritis.
  Class IIB: there is severe intimal arteritis comprising at least 25% of the lumenal area.
  Class III: there is transmural (e.g. the full vessel wall thickness) arteritis.
Time Frame: 3, 6 and 12 months post transplant
Measure: Number; unit: participants
Arm/Group | Myfortic Preload | Myfortic Standard
Number analyzed (Participants) | 40 | 21
participants
  3 months | 7 | 3
  6 months | 7 | 3
  12 months | 8 | 4

2. Secondary Outcome: Severity of Acute Rejection by Banff '97 Criteria
Description: Severity of biopsy-confirmed acute rejection by Banff '97 Criteria (updated 2007) at 1 year. The acute form of T-cell mediated rejection is furthermore subclassified as follows. Since this is the most common form of rejection, it is useful to know:
  As with humoral rejection, there are both acute & chronic forms:
  The acute form of T-cell mediated rejection is furthermore subclassified as follows. Since this is the most common form of rejection, it is useful to know:
  Class IA: there is at least 25% of parenchymal showing interstitial infiltration and foci of moderate tubulitis (defined as a certain number of immune cells present in tubular cross-sections).
  Class IB: just like Class IA except there is more severe tubulitis.
  Class IIA: there is mild-to-moderate intimal arteritis.
  Class IIB: there is severe intimal arteritis comprising at least 25% of the lumenal area.
  Class III: there is transmural (e.g. the full vessel wall thickness) arteritis.
Time Frame: Severity 1 year post transplant
Measure: Number; unit: participants
Arm/Group | Myfortic Preload | Myfortic Standard
Number analyzed (Participants) | 40 | 21
participants
  Grade IA | 3 | 1
  Grade IB | 4 | 1
  Grade IIA | 1 | 0
  Grade IIB | 0 | 0
  Antibody Mediated Rejection | 0 | 1
  Mixed Acute Rejection | 0 | 1

3. Secondary Outcome: Difference in Renal Function
Description: Difference in renal function between groups at listed time points assessed by mean serum creatinine. Increased serum creatinine could indicate worsening renal function. A "normal" serum creatinine range for the transplant population varies by patient, but a typical range for Scr would be 1-2 mg/dL.
Time Frame: Difference at 1 month, 3 months, 6 months, 1 year
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Myfortic Preload | Myfortic Standard
Number analyzed (Participants) | 40 | 21
mg/L
  1 month | 1.41 (0.4) | 1.43 (0.6)
  3 months | 1.45 (0.5) | 1.39 (0.5)
  6 months | 1.43 (0.4) | 1.40 (0.6)
  1 year | 1.36 (0.4) | 1.5 (1.0)

4. Secondary Outcome: Incidence of Chronic Alloantibody Rejection or Chronic Allograft Arteriopathy by Banff '97
Description: The Banff features suggestive of chronic rejection were: a) chronic transplant glomerulopathy: Glomerular basement membrane duplication and mesangial cell proliferation, and b) vasculopathy: Fibrous intimal thickening often with fragmentation of internal elastic lamina. Chronic changes in the interstitium (ci), tubules (ct), vessels (cv), and glomerulus (cg) were likewise graded into 0, 1, 2, and 3. The severity of interstitial fibrosis and tubular atrophy, as also chronic transplant glomerulopathy and vasculopathy were used to grade chronic allograft changes.
Time Frame: 1 year
Measure: Number; unit: participants
Arm/Group | Myfortic Preload | Myfortic Standard
Number analyzed (Participants) | 40 | 21
participants
  mild Chronic allograft nephropathy (CAN) | 9 | 3
  Moderate Chronic allograft nephropathy (CAN) | 0 | 1

5. Secondary Outcome: Number of Patients Requiring Anti-lymphocyte Therapy for Acute Rejection
Time Frame: 1 year
Measure: Number; unit: participants
Arm/Group | Myfortic Preload | Myfortic Standard
Number analyzed (Participants) | 40 | 21
participants
  Pulse methylprednisolone | 5 | 3
  Thymoglobulin | 6 | 0
  Plasmapheresis | 0 | 2
  Intravenous immunoglobulin (IVIg) | 0 | 0
  Rituximab | 0 | 1

ADVERSE EVENTS:
Arm/Group | Myfortic Preload | Myfortic Standard
Serious Adverse Events (participants affected / at risk) | 19/40 | 10/21
Other Adverse Events (participants affected / at risk) | 14/40 | 8/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Myfortic Preload (N=40) | Myfortic Standard (N=21)
Purcutaneous Nephrostomy (Renal and urinary disorders) | 0 (0) | 1 (1)
Borderline Rejection (Renal and urinary disorders) | 3 (3) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Renal Dysfunction (Renal and urinary disorders) | 5 (6) | 3 (4)
Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Small Bowel Obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Fluid Aspiration (Renal and urinary disorders) | 1 (1) | 0 (0)
Acute Hypoxemic Respiration Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Slow Creatine Decline (Renal and urinary disorders) | 1 (1) | 0 (0)
Wound Incision Infection (Infections and infestations) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 4 (4) | 2 (2)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 1 (3)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 4 (4) | 2 (4)
Vomiting (Gastrointestinal disorders) | 4 (4) | 3 (3)
Acute Allograft Dysfunction (Renal and urinary disorders) | 0 (0) | 1 (1)
Fever (General disorders) | 2 (2) | 2 (2)
Left Internal Carotid Artery Stenosis (Cardiac disorders) | 0 (0) | 1 (1)
Hyperkalemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Gout Imflammation (General disorders) | 1 (1) | 0 (0)
Serum Creatinine Increased (Renal and urinary disorders) | 6 (12) | 4 (7)
E Coli Bactermia (Infections and infestations) | 1 (1) | 0 (0)
Rebabilitation of Debility (General disorders) | 1 (1) | 0 (0)
Chest Pain (Cardiac disorders) | 1 (1) | 0 (0)
Acute Mediated Rejection (Renal and urinary disorders) | 0 (0) | 1 (3)
Impotence (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Erectile Dysfunction (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Bicarbonate Decrease (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Metabolic Acidosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
High Blood Sugar (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 3 (3) | 0 (0)
Ureteral Revision (Renal and urinary disorders) | 1 (1) | 0 (0)
Banff 2A Rejection (Renal and urinary disorders) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Elevated Liver Enzymes (Hepatobiliary disorders) | 1 (1) | 0 (0)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Elevated Postassium (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Obstructive Uropathy (Renal and urinary disorders) | 1 (1) | 0 (0)
Wound Dehiscense (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
BK Virus (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Perinephric Lymphocele (Renal and urinary disorders) | 1 (1) | 1 (1)
Urothelial Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Urinary Tract Infection (Renal and urinary disorders) | 0 (0) | 1 (1)
Disseminated Histoplasmosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Myfortic Preload (N=40) | Myfortic Standard (N=21)
Headache (General disorders) | 1 (1) | 0 (0)
Dizziness (General disorders) | 1 (1) | 0 (0)
Weight Loss (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Cytomegalovirus (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 1 (3)
Diarrhea (Gastrointestinal disorders) | 4 (4) | 4
Vomiting (Gastrointestinal disorders) | 4 | 3 (3)
Nausea (Gastrointestinal disorders) | 6 | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No